CLINICAL TRIAL: NCT00397150
Title: PROMISE EBF: Promoting Infant Health and Nutrition in Sub-Saharan Africa: Safety and Efficacy of Exclusive Breastfeeding Promotion in the Era of HIV
Brief Title: PROMISE EBF: Safety and Efficacy of Exclusive Breastfeeding Promotion in the Era of HIV in Sub-Saharan Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre For International Health (Other)
Collaborators: European Union (Other); The Norwegian Programme for Development, Research and Higher Education (Other); University of Bergen (Other); Université Montpellier (Other); Uppsala University (Other); Centre Muraz (Other); Makerere University (Other); University of Zambia (Other); University of the Western Cape (Other)
Responsible Party: Principal Investigator, Thorkild Tylleskar, Professor, Centre For International Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: INCO-CT-2004-003660
Record Dates: First submitted 2006-11-07; First posted 2006-11-08 (Estimated); Results first posted 2015-02-24 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-02

CONDITIONS: Diarrhea
Keywords: Infant Nutrition [G06.696.259.750]; Infant Care [N02.421.088.120] +; Diarrhea, Infantile [C23.888.821.214.500]; Child Health Services [N02.421.143.130] +; Counseling [N02.421.143.303]; Growth [G07.574.249] +; Micronutrients [D11.430]; Breast Feeding [G06.696.259.750.500]
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Peer-support for exclusive breastfeeding
  Interventions: Behavioral: Peer-support for exclusive breastfeeding
- No intervention (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Peer-support for exclusive breastfeeding — Counselling to support exclusive breastfeeding up to the age of 6 months of age by the use of peer-counsellors in the local community
  Arms: Intervention

SUMMARY:
The objective of the project is to develop and test an intervention to promote exclusive breastfeeding (EBF), to assess its impact on infant health in African contexts where a high prevalence of HIV is a barrier, and to strengthen the evidence base regarding the optimal duration for EBF.

Promotion of EBF is the most effective child health intervention currently feasible for implementation at the population level in low-income countries. It can lower infant mortality by 13%, and by an additional 2% were it not for the fact that breastfeeding transmits HIV. Only recently proven to be possible in hot and even dry climates, EBF without even offering water is still little appreciated by mothers or supported by health workers. EBF rates are especially low in Africa but the potential for rapid implementation may be high. A few studies elsewhere suggest that peer counselling can often achieve dramatic increases. Thus the investigators will run the first randomised trial to develop and test models for applying this approach in four African countries and to quantify health benefits, cost-effectiveness, and implications for the health care system.

While experts realize that the HIV threat ought not to present much of a biological constraint to promoting EBF, in heavily affected countries it does represent a cultural constraint. Overcoming this will require the development of a safe and effective means of promoting EBF that is HIV-sensitive by taking into account the need to minimise postnatal HIV transmission.

Another scientific constraint to the promotion of exclusive breastfeeding for six months, as recommended by the World Health Organization (WHO), is uncertainty about its impact on the micronutrient status of infants. In a substudy, the investigators will carefully follow markers of infant micronutrient status to see how they vary by feeding pattern, including EBF, for a longer period than has been examined previously.

DETAILED DESCRIPTION:
Rationale

The single most effective way of saving the lives of millions of young children in developing countries would be the promotion of exclusive breastfeeding (EBF). Over a period of 10 years it could save the lives of an estimated 15 million children.

"Infants aged 0-5 months who are not breastfed have seven-fold and five-fold increased risks of death from diarrhoea and pneumonia respectively, compared with infants who are exclusively breastfed. At the same age, non-exclusive rather than exclusive breastfeeding results in more than two-fold increased risks of dying from diarrhoea and pneumonia." Lancet 2003; 361: 2226-34

This assertion, and related comments and findings, set out by the Bellagio Child Survival Group in a recent article in the Lancet summarising findings from international research of how best to reduce infant mortality in developing countries, is made despite our limited knowledge of how best to promote EBF. This proposal addresses the urgent need to tackle this limitation. How best to promote EBF needs attention because it will be necessary to secure high rates of support for EBF from young mothers, and we do not currently know the best way to bring this about, particularly in the cultural context of Africa. Unless we can find more effective strategies to combat poor feeding practices in both health facility and community settings, the child mortality rate will continue to be high.

Breastfeeding

The benefits of breastfeeding and the negative effects of artificial feeding in underprivileged environments were clearly brought to the public attention in the 1970s, backed by increasingly strong scientific support. As a result the International Code of Marketing of Breast-milk Substitutes and subsequent World Health Assembly Resolutions were created in the 1980s to avoid the marketing of infant foods, teats and bottles in ways that could interfere with breastfeeding. In the early 1990s, UNICEF started the "Baby-friendly Hospital Initiative" (BFHI), which decreased many of the practices in the health care system that had a negative impact on breastfeeding. Together with many of the other child health programmes during these decades these interventions contributed to a reduction in child morbidity and mortality.

Exclusive Breastfeeding - An Even Better Version of Breastfeeding

EBF means that the infant receives nothing else other than breast milk, not even water. That breastfed children do not need anything besides breast milk, not even water, and not even in hot climates, was discovered in the 1970s. A decade of research confirmed this, followed by an attempt to define breastfeeding into various patterns by WHO.

EBF is not a traditional concept; beliefs and practices regarding a wide range of early supplements are common around the world, and often seem to reflect beliefs expressed by early physicians. Nor is it widely understood by health care professionals, given the lack of information on it even in most paediatric basic training.

So if EBF is able to lower child mortality by 13%, why is it not promoted on a large scale already today? Two major reasons are: fear of HIV transmission through breast milk and uncertainty about the micronutrient status in children exclusively breastfed for 6 months.

Breastfeeding and Risk of HIV Transmission

When an HIV-positive mother breastfeeds for 1.5 years or more, this appears to lead to an additional 15% risk of postnatal HIV transmission on average. At a population level the epidemiological evidence is that exclusive breastfeeding should still be promoted even in countries with a high prevalence of HIV. For many HIV positive mothers the risk of transmitting HIV to their children is outweighed by the risk of the infant dying if not breastfed because of the poor socioeconomic and environmental conditions they live in. Limited evidence suggests that for these women and their children EBF is even more important, not just for minimising respiratory and gastrointestinal infections but also perhaps in reducing the risk of HIV transmission. However in reality the HIV epidemic has undermined breastfeeding promotion efforts especially in countries that would benefit the most. In addition, expensive approaches of dealing with HIV have removed the focus from breastfeeding as an inexpensive way of promoting optimal child health.

Intervention: Peer Counselling

The constraints discussed above have meant that efforts to promote EBF have been rudimentary so far, consisting mainly of the Baby-Friendly Hospital Initiative. But in Africa nearly all such efforts have come almost to a complete standstill in recent years. EBF promotion therefore needs to be reshaped in this era of HIV. The challenge is to urgently put back on track the promotion of exclusive breastfeeding for the benefit of the world's children without losing credibility by doing it indiscriminately. PROMISE will fine-tune and test an upgraded version of EBF-promotion that is HIV-sensitive and do it in four African countries with a high prevalence of HIV where it is most needed. In particular, it will be the first study to deal explicitly with each of these constraints, opening the way for a more widespread and successful promotion of EBF, especially in Africa, ultimately giving back to Africa one of the powerful and cheap interventions to prevent child mortality and morbidity.

Peer counselling is a proven cost-effective approach for changing behaviour, for example, preventing HIV infection. Several studies have also examined its impact on breastfeeding behaviour. Based largely on quasi-experimental studies peer counselling was shown to have an impact on the duration of any breastfeeding.

Potential Impact

This study will provide the first data from a randomised trial on the safety and efficacy of peer counselling as a way of increasing rates of exclusive breastfeeding in the African context. Outcomes include morbidity, growth, and micronutrient status.

PROMISE EBF will provide an example to the world of how efforts to promote exclusive breastfeeding and avoid postnatal HIV transmission can be done jointly, and what synergisms may result. Methods employed and costs will be documented and reported on to increase the ease of replication and sustainability.

In Africa, there is a growing awareness that strategies must be identified and tested that can lead to the highest possible infant survival rate in the face of the risk of postnatal HIV transmission. In 1997 UNAIDS, WHO and UNICEF changed their policy on HIV and infant feeding, and issued guidelines for implementing this new policy a year later. Whereas previously countries where most infant mortality was due to infection and malnutrition were advised to promote breastfeeding irrespective of the mother's HIV status, the new policy called for individual counselling on the advantages and disadvantages of breastfeeding vs. artificial feeding that would enable mothers to make an informed choice. UNICEF provided free formula at a number of pilot sites.

Methodology

Design

A prospective, multi-center, community-randomised, controlled, experimental design will be used to execute this trial.

Randomization

A number of over 30 randomisation units should be identified within a reasonable distance from the study office. The randomisation unit varies between sites but will typically be 1-2 villages with an average of 1000 inhabitants (about 35 infants born per year given a birth rate of 3%). Before engaging in the selection of communities, extensive information will be given to community leaders and the rest of the selection process will be done in close collaboration with community leaders. Within the district the suitable communities will be selected and groups considered similar, based on location, urban-rural, and socioeconomic status will be stratified. Care will be taken to allow for 'corridors' between selected communities to be randomised. In each stratum half of the communities will be randomised to intervention and the reminder to control communities. Local community leaders will be further informed about the study.

Each of the clusters should be visited and checked for size, for collaborative administrative leaders, and for not sharing important facilities (water supply, market/shop/trading centre, primary school, mosque, church) with any other potential cluster. If both urban and rural clusters are included no less than 30% of each should be included. The complete list of randomisable clusters will be checked and 24 clusters will be randomised in each site, if applicable in the rural/urban strata.

The study will be carried out in four African countries, Burkina Faso in French-speaking West Africa, Uganda in East Africa, Zambia in Central Africa and South Africa in Southern Africa.

In each country one or more districts have been selected as the intervention sites, Banfora in the South-west of Burkina-Faso, Mbale District in Eastern Uganda, Mazabuka in Southern Province in Zambia and three sites in South Africa: Umlazi in Durban, KwaZulu Natal, Rietvlei in the Eastern Cape and Paarl in the Western Cape. Pregnant women in the randomised communities (= clusters) will be informed about the study and asked if they are willing to participate. If they agree, an enrolment interview will be carried out and based on eligibility criteria the women will or will not be accepted into the study.

Sample Size and Power

Of the primary outcome measures the decrease in diarrhoea is the most difficult to catch. We have based our sample size calculation on the expected reduction in cases of diarrhoea (at the age of 3 months) over the last two weeks of one third from 12% to 8%. With a 95% confidence interval (alpha error 0.05) and power of 80%, an average number of infants of 35 per randomised community, and a coefficient of variation between the communities of 0.3, we will need to randomise 48 communities in each arm - a total of 96 communities. This will include 420 infants in each arm in each country, a total of 840 children per country and all in all 3360 children studied across the four sites. This sample size will very accurately give us the increase in EBF and be able to document the above decrease in diarrhoea morbidity.

Recruitment Procedure

The recruitment procedure will be adapted to the local circumstances. In the most common case, each cluster will have a recruiter ("pregnancy monitor") who will be a mature woman of good repute living within the cluster. The pregnancy monitors will inform the research centre about pregnant women that may be eligible to participate in the study. A data collector/research assistant will be sent to visit the woman to ascertain eligibility, obtain consent to participate in the study and conduct the recruitment interview.

In South Africa, the recruitment of women will be done at the health facility in the antenatal clinic, where a data collector/research assistant will interview the woman to ascertain eligibility, obtain consent to participate in the study and conduct the recruitment interview.

ELIGIBILITY:
Inclusion Criteria:

* Lives in a selected cluster
* Is >= 6 months pregnant
* Has no plans to move outside of the cluster within 1 year

Exclusion Criteria:

* Reduced ability to collaborate for psychological/mental reasons
* Severely ill
* Has given birth more than 7 days ago
* Has given birth less than 7 days ago and it was a multiple birth; or the child has a severe malformation; or death of the mother or the baby.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2579 (Actual)
Dates: Start 2006-11; Primary Completion 2008-07 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thorkild Tylleskar, MD, PHD, Principal Investigator — Centre For International Health
Locations (4):
- Centre Muraz, Bobo-Dioulasso, Burkina Faso
- School of Public Health, University of the Western Cape (UWC), Cape Town, South Africa
- Dept of Paediatrics and Child Health, Makerere University, Kampala, Uganda
- Dept of Paediatrics and Child Health, University of Zambia, School of Medicine (UNZA/SOM), Lusaka, Zambia

REFERENCES:
- [Background] Fadnes LT, Nankabirwa V, Sommerfelt H, Tylleskar T, Tumwine JK, Engebretsen IM; PROMISE-EBF Study Group. Is vaccination coverage a good indicator of age-appropriate vaccination? A prospective study from Uganda. Vaccine. 2011 Apr 27;29(19):3564-70. doi: 10.1016/j.vaccine.2011.02.093. Epub 2011 Mar 12. PMID 21402043
- [Background] Nankabirwa V, Tylleskar T, Tumwine JK, Sommerfelt H; Promise-ebf Study Group. Maternal education is associated with vaccination status of infants less than 6 months in Eastern Uganda: a cohort study. BMC Pediatr. 2010 Dec 15;10:92. doi: 10.1186/1471-2431-10-92. PMID 21159193
- [Background] Nkonki LL, Daniels KL; PROMISE-EBF study group. Selling a service: experiences of peer supporters while promoting exclusive infant feeding in three sites in South Africa. Int Breastfeed J. 2010 Oct 26;5:17. doi: 10.1186/1746-4358-5-17. PMID 20977716
- [Background] Nankunda J, Tumwine JK, Nankabirwa V, Tylleskar T; PROMISE-EBF Study Group. "She would sit with me": mothers' experiences of individual peer support for exclusive breastfeeding in Uganda. Int Breastfeed J. 2010 Oct 26;5:16. doi: 10.1186/1746-4358-5-16. PMID 20977715
- [Background] Engebretsen IM, Moland KM, Nankunda J, Karamagi CA, Tylleskar T, Tumwine JK. Gendered perceptions on infant feeding in Eastern Uganda: continued need for exclusive breastfeeding support. Int Breastfeed J. 2010 Oct 26;5:13. doi: 10.1186/1746-4358-5-13. PMID 20977712
- [Background] Engebretsen IM, Shanmugam R, Sommerfelt AE, Tumwine JK, Tylleskar T. Infant feeding modalities addressed in two different ways in Eastern Uganda. Int Breastfeed J. 2010 Feb 4;5(1):2. doi: 10.1186/1746-4358-5-2. PMID 20205864
- [Background] Wandera MN, Engebretsen IM, Rwenyonyi CM, Tumwine J, Astrom AN; PROMISE-EBF Study Group. Periodontal status, tooth loss and self-reported periodontal problems effects on oral impacts on daily performances, OIDP, in pregnant women in Uganda: a cross-sectional study. Health Qual Life Outcomes. 2009 Oct 14;7:89. doi: 10.1186/1477-7525-7-89. PMID 19828031
- [Background] Nor B, Zembe Y, Daniels K, Doherty T, Jackson D, Ahlberg BM, Ekstrom EC; PROMISE-EBF Study Group. "Peer but not peer": considering the context of infant feeding peer counseling in a high HIV prevalence area. J Hum Lact. 2009 Nov;25(4):427-34. doi: 10.1177/0890334409341050. Epub 2009 Jul 21. PMID 19622755
- [Background] Wandera M, Engebretsen IM, Okullo I, Tumwine JK, Astrom AN; PROMISE-EBF Study Group. Socio-demographic factors related to periodontal status and tooth loss of pregnant women in Mbale district, Uganda. BMC Oral Health. 2009 Jul 18;9:18. doi: 10.1186/1472-6831-9-18. PMID 19615094
- [Background] Fjeld E, Siziya S, Katepa-Bwalya M, Kankasa C, Moland KM, Tylleskar T; PROMISE-EBF Study Group. 'No sister, the breast alone is not enough for my baby' a qualitative assessment of potentials and barriers in the promotion of exclusive breastfeeding in southern Zambia. Int Breastfeed J. 2008 Nov 5;3:26. doi: 10.1186/1746-4358-3-26. PMID 18986539
- [Background] Daniels K, Nor B, Jackson D, Ekstrom EC, Doherty T. Supervision of community peer counsellors for infant feeding in South Africa: an exploratory qualitative study. Hum Resour Health. 2010 Mar 30;8:6. doi: 10.1186/1478-4491-8-6. PMID 20353561
- [Background] Fadnes LT, Engebretsen IM, Moland KM, Nankunda J, Tumwine JK, Tylleskar T. Infant feeding counselling in Uganda in a changing environment with focus on the general population and HIV-positive mothers - a mixed method approach. BMC Health Serv Res. 2010 Sep 6;10:260. doi: 10.1186/1472-6963-10-260. PMID 20815932
- [Background] Engebretsen IM, Wamani H, Karamagi C, Semiyaga N, Tumwine J, Tylleskar T. Low adherence to exclusive breastfeeding in Eastern Uganda: a community-based cross-sectional study comparing dietary recall since birth with 24-hour recall. BMC Pediatr. 2007 Mar 1;7:10. doi: 10.1186/1471-2431-7-10. PMID 17331251
- [Background] Engebretsen IM, Tylleskar T, Wamani H, Karamagi C, Tumwine JK. Determinants of infant growth in Eastern Uganda: a community-based cross-sectional study. BMC Public Health. 2008 Dec 22;8:418. doi: 10.1186/1471-2458-8-418. PMID 19102755
- [Background] Fadnes LT, Engebretsen IM, Wamani H, Wangisi J, Tumwine JK, Tylleskar T. Need to optimise infant feeding counselling: a cross-sectional survey among HIV-positive mothers in Eastern Uganda. BMC Pediatr. 2009 Jan 9;9:2. doi: 10.1186/1471-2431-9-2. PMID 19134187
- [Background] Fadnes LT, Engebretsen IM, Wamani H, Semiyaga NB, Tylleskar T, Tumwine JK. Infant feeding among HIV-positive mothers and the general population mothers: comparison of two cross-sectional surveys in Eastern Uganda. BMC Public Health. 2009 May 7;9:124. doi: 10.1186/1471-2458-9-124. PMID 19422709
- [Background] Nankunda J, Tylleskar T, Ndeezi G, Semiyaga N, Tumwine JK; PROMISE-EBF Study Group. Establishing individual peer counselling for exclusive breastfeeding in Uganda: implications for scaling-up. Matern Child Nutr. 2010 Jan;6(1):53-66. doi: 10.1111/j.1740-8709.2009.00187.x. PMID 20055930
- [Background] Nankunda J, Tumwine JK, Soltvedt A, Semiyaga N, Ndeezi G, Tylleskar T. Community based peer counsellors for support of exclusive breastfeeding: experiences from rural Uganda. Int Breastfeed J. 2006 Oct 20;1:19. doi: 10.1186/1746-4358-1-19. PMID 17054796
- [Background] Fadnes LT, Jackson D, Engebretsen IM, Zembe W, Sanders D, Sommerfelt H, Tylleskar T; PROMISE-EBF Study Group. Vaccination coverage and timeliness in three South African areas: a prospective study. BMC Public Health. 2011 May 27;11:404. doi: 10.1186/1471-2458-11-404. PMID 21619642
- [Background] Ramokolo V, Lombard C, Fadnes LT, Doherty T, Jackson DJ, Goga AE, Chhagan M, Van den Broeck J. HIV infection, viral load, low birth weight, and nevirapine are independent influences on growth velocity in HIV-exposed South African infants. J Nutr. 2014 Jan;144(1):42-8. doi: 10.3945/jn.113.178616. Epub 2013 Nov 6. PMID 24198309
- [Result] Diallo AH, Meda N, Zabsonre E, Sommerfelt H, Cousens S, Tylleskar T; PROMISE-EBF Study Group. Perinatal mortality in rural Burkina Faso: a prospective community-based cohort study. BMC Pregnancy Childbirth. 2010 Aug 17;10:45. doi: 10.1186/1471-2393-10-45. PMID 20716352
- [Result] Diallo AH, Meda N, Ouedraogo WT, Cousens S, Tylleskar T; PROMISE-EBF Study Group. A prospective study on neonatal mortality and its predictors in a rural area in Burkina Faso: can MDG-4 be met by 2015? J Perinatol. 2011 Oct;31(10):656-63. doi: 10.1038/jp.2011.6. Epub 2011 Mar 3. PMID 21372798
- [Result] Tylleskar T, Jackson D, Meda N, Engebretsen IM, Chopra M, Diallo AH, Doherty T, Ekstrom EC, Fadnes LT, Goga A, Kankasa C, Klungsoyr JI, Lombard C, Nankabirwa V, Nankunda JK, Van de Perre P, Sanders D, Shanmugam R, Sommerfelt H, Wamani H, Tumwine JK; PROMISE-EBF Study Group. Exclusive breastfeeding promotion by peer counsellors in sub-Saharan Africa (PROMISE-EBF): a cluster-randomised trial. Lancet. 2011 Jul 30;378(9789):420-7. doi: 10.1016/S0140-6736(11)60738-1. PMID 21752462
- [Result] Nankabirwa V, Tylleskar T, Nankunda J, Engebretsen IM, Sommerfelt H, Tumwine JK; PROMISE EBF Research Consortium. Malaria parasitaemia among infants and its association with breastfeeding peer counselling and vitamin A supplementation: a secondary analysis of a cluster randomized trial. PLoS One. 2011;6(7):e21862. doi: 10.1371/journal.pone.0021862. Epub 2011 Jul 7. PMID 21760916
- [Result] Nankabirwa V, Tumwine JK, Tylleskar T, Nankunda J, Sommerfelt H; PROMISE EBF Research Consortium. Perinatal mortality in eastern Uganda: a community based prospective cohort study. PLoS One. 2011 May 9;6(5):e19674. doi: 10.1371/journal.pone.0019674. PMID 21573019
- [Result] Chola L, Fadnes LT, Engebretsen IM, Tumwine JK, Tylleskar T, Robberstad B; PROMISE EBF Study Group. Infant feeding survival and Markov transition probabilities among children under age 6 months in Uganda. Am J Epidemiol. 2013 Mar 1;177(5):453-62. doi: 10.1093/aje/kws254. Epub 2013 Feb 5. PMID 23384876
- [Result] Nkonki LL, Daviaud E, Jackson D, Chola L, Doherty T, Chopra M, Robberstad B; Promise-EBF Study Group. Costs of promoting exclusive breastfeeding at community level in three sites in South Africa. PLoS One. 2014 Jan 10;9(1):e79784. doi: 10.1371/journal.pone.0079784. eCollection 2014. PMID 24427264
- [Result] Engebretsen IM, Jackson D, Fadnes LT, Nankabirwa V, Diallo AH, Doherty T, Lombard C, Swanvelder S, Nankunda J, Ramokolo V, Sanders D, Wamani H, Meda N, Tumwine JK, Ekstrom EC, Van de Perre P, Kankasa C, Sommerfelt H, Tylleskar T; PROMISE EBF-study group. Growth effects of exclusive breastfeeding promotion by peer counsellors in sub-Saharan Africa: the cluster-randomised PROMISE EBF trial. BMC Public Health. 2014 Jun 21;14:633. doi: 10.1186/1471-2458-14-633. PMID 24950759
- [Result] Doherty T, Jackson D, Swanevelder S, Lombard C, Engebretsen IM, Tylleskar T, Goga A, Ekstrom EC, Sanders D; PROMISE EBF study group. Severe events in the first 6 months of life in a cohort of HIV-unexposed infants from South Africa: effects of low birthweight and breastfeeding status. Trop Med Int Health. 2014 Oct;19(10):1162-9. doi: 10.1111/tmi.12355. Epub 2014 Jul 23. PMID 25053420
- [Derived] Birungi N, Fadnes LT, Kasangaki A, Nankabirwa V, Okullo I, Lie SA, Tumwine JK, Astrom AN; PROMISE-EBF study group. Assessing causal effects of early life-course factors on early childhood caries in 5-year-old Ugandan children using directed acyclic graphs (DAGs): A prospective cohort study. Community Dent Oral Epidemiol. 2017 Dec;45(6):512-521. doi: 10.1111/cdoe.12314. Epub 2017 Jun 20. PMID 28631283
- [Derived] Eide KT, Fadnes LT, Engebretsen IM, Onarheim KH, Wamani H, Tumwine JK, Norheim OF; PROMISE-EBF Study Group. Impact of a peer-counseling intervention on breastfeeding practices in different socioeconomic strata: results from the equity analysis of the PROMISE-EBF trial in Uganda. Glob Health Action. 2016 Jul 28;9:30578. doi: 10.3402/gha.v9.30578. eCollection 2016. PMID 27473676
- [Derived] Fadnes LT, Nankabirwa V, Engebretsen IM, Sommerfelt H, Birungi N, Lombard C, Swanevelder S, Van den Broeck J, Tylleskar T, Tumwine JK; PROMISE-EBF Study Group. Effects of an exclusive breastfeeding intervention for six months on growth patterns of 4-5 year old children in Uganda: the cluster-randomised PROMISE EBF trial. BMC Public Health. 2016 Jul 12;16:555. doi: 10.1186/s12889-016-3234-3. PMID 27405396
- [Derived] Birungi N, Fadnes LT, Okullo I, Kasangaki A, Nankabirwa V, Ndeezi G, Tumwine JK, Tylleskar T, Lie SA, Astrom AN. Effect of Breastfeeding Promotion on Early Childhood Caries and Breastfeeding Duration among 5 Year Old Children in Eastern Uganda: A Cluster Randomized Trial. PLoS One. 2015 May 4;10(5):e0125352. doi: 10.1371/journal.pone.0125352. eCollection 2015. PMID 25938681
- [Derived] Engebretsen IM, Nankabirwa V, Doherty T, Diallo AH, Nankunda J, Fadnes LT, Ekstrom EC, Ramokolo V, Meda N, Sommerfelt H, Jackson D, Tylleskar T, Tumwine JK; PROMISE-EBF study group. Early infant feeding practices in three African countries: the PROMISE-EBF trial promoting exclusive breastfeeding by peer counsellors. Int Breastfeed J. 2014 Nov 18;9:19. doi: 10.1186/1746-4358-9-19. eCollection 2014. PMID 25784955
- [Derived] Zembe-Mkabile W, Doherty T, Sanders D, Jackson D, Chopra M, Swanevelder S, Lombard C, Surender R. Why do families still not receive the child support grant in South Africa? A longitudinal analysis of a cohort of families across South Africa. BMC Int Health Hum Rights. 2012 Oct 22;12:24. doi: 10.1186/1472-698X-12-24. PMID 23088827
- [Derived] Hama Diallo A, Meda N, Sommerfelt H, Traore GS, Cousens S, Tylleskar T; PROMISE-EBF Study Group. The high burden of infant deaths in rural Burkina Faso: a prospective community-based cohort study. BMC Public Health. 2012 Sep 5;12:739. doi: 10.1186/1471-2458-12-739. PMID 22947029
- [Derived] Doherty T, Sanders D, Jackson D, Swanevelder S, Lombard C, Zembe W, Chopra M, Goga A, Colvin M, Fadnes LT, Engebretsen IM, Ekstrom EC, Tylleskar T; PROMISE EBF study group. Early cessation of breastfeeding amongst women in South Africa: an area needing urgent attention to improve child health. BMC Pediatr. 2012 Jul 24;12:105. doi: 10.1186/1471-2431-12-105. PMID 22827969
- See also: Centre for International Health, University of Bergen, Norway — http://www.uib.no/cih/en

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pregnant women are recruited in their communities.
Groups:
- Intervention: Peer-counselling for exclusive breastfeeding
- No Intervention: Standard of care
Period: Overall Study
Arm/Group | Intervention | No Intervention
Started | 1323 | 1256
Completed | 1188 | 1111
Not Completed | 135 | 145

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | No Intervention | Total
Number analyzed (Participants) | 1323 | 1256 | 2579
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1323 | 1256 | 2579
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: days] | 7 [5 to 9] | 7 [5 to 9] | 7 [5 to 9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 662 | 628 | 1290
  Male | 661 | 628 | 1289
Region of Enrollment [Number; unit: participants]
  Burkina Faso | 392 | 402 | 794
  Uganda | 396 | 369 | 765
  South Africa | 535 | 485 | 1020

OUTCOME MEASURES:

1. Primary Outcome: Exclusive Breastfeeding Rates in Burkina Faso
Description: The EBF prevalences (24-h recall) at 12 weeks in the intervention and control clusters.
Time Frame: at 3 months of age
Population: ITT
Measure: Number; unit: participants
Arm/Group | Intervention | No Intervention
Number analyzed (Participants) | 392 | 402
participants | 310 | 161
Statistical Analysis 1: Comparison: Intervention vs No Intervention; Test type: Superiority or Other; Prevalence ratio = 2.29, 95% CI 2-sided [1.33 to 3.92]

2. Primary Outcome: Infant Morbidity, 2 Week Diarrhoea Prevalence
Time Frame: at 3 months of age
Measure: Number; unit: participants
Arm/Group | Intervention | No Intervention
Number analyzed (Participants) | 1323 | 1256
participants | 104 | 101

3. Secondary Outcome: Growth
Time Frame: (up to 6 months of age)
Reporting Status: Not Posted

4. Secondary Outcome: Per Protocol Analysis of EBF Rates
Time Frame: at 3 months of age
Reporting Status: Not Posted

5. Secondary Outcome: Per Protocol Analysis of Infant Morbidity
Time Frame: at 3 months of age
Reporting Status: Not Posted

6. Primary Outcome: Exclusive Breastfeeding Rates in Uganda
Description: The EBF prevalences (24-h recall) at 12 weeks in the intervention and control clusters.
Time Frame: at 3 months of age
Population: ITT
Measure: Number; unit: participants
Arm/Group | Intervention | No Intervention
Number analyzed (Participants) | 396 | 369
participants | 323 | 161
Statistical Analysis 1: Comparison: Intervention vs No Intervention; Test type: Superiority or Other; Prevalence ratio = 1.89, 95% CI 2-sided [1.70 to 2.11]

7. Primary Outcome: Exclusive Breastfeeding Rates in South Africa
Description: The EBF prevalences based on 24-h recall at 12 weeks in the intervention and control clusters.
Time Frame: at 3 months of age
Population: ITT
Measure: Number; unit: participants
Arm/Group | Intervention | No Intervention
Number analyzed (Participants) | 535 | 485
participants | 56 | 30
Statistical Analysis 1: Comparison: Intervention vs No Intervention; Test type: Superiority or Other; Prevalence ratio = 1.72, 95% CI 2-sided [1.12 to 2.63]

ADVERSE EVENTS:
Arm/Group | Peer Counselling for Exclusive Breastfeeding | Standard of Care
Serious Adverse Events (participants affected / at risk) | 32/1323 | 22/1256
Other Adverse Events (participants affected / at risk) | 0/1323 | 0/1256
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peer Counselling for Exclusive Breastfeeding (N=1323) | Standard of Care (N=1256)
Death (Infections and infestations) | 32 (32) | 22 (22)

LIMITATIONS AND CAVEATS:
Trial not entirely blinded.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No